CLINICAL TRIAL: NCT01199198
Title: Randomized Placebo-Controlled Trial of Tolvaptan in Hyponatremic Patients With Cancer
Brief Title: Tolvaptan in Hyponatremic Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-0862
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Advanced Cancers
Keywords: Hyponatremia; Serum sodium; Tolvaptan; Placebo
MeSH Terms: conditions — Hyponatremia | interventions — Tolvaptan; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan Group (Experimental): Tolvaptan Group: Starting dose 15 mg by mouth once a day for 14 days.
  Interventions: Drug: Tolvaptan
- Placebo Group (Placebo Comparator): Placebo Group: Placebo by mouth once a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — Starting dose 15 mg by mouth once a day for 14 days.
  Other Names: Samsca
  Arms: Tolvaptan Group
Drug: Placebo — Placebo by mouth once a day for 14 days.
  Other Names: Sugar Pill
  Arms: Placebo Group

SUMMARY:
The goal of this clinical research study is to learn if tolvaptan can help raise salt (sodium) levels in the cancer patients' blood by removing extra body water as urine.

DETAILED DESCRIPTION:
The Study Drug:

Tolvaptan is designed to help raise salt levels in your blood by removing extra body water as urine.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being assigned to either group:

* If you are in Group 1, you will take tolvaptan and receive standard of care
* If you are in Group 2, you will take a placebo and receive the standard of care for patients with hyponatremia. A placebo is a tablet that looks like the study drug but has no active ingredients.

You will not know which group you are assigned. However, if needed for your safety, you will be able to find out what you are receiving at any time.

Study Drug Administration:

You will take tolvaptan or the placebo 1 time every day by mouth for 14 days.

If you are receiving the placebo, you will also receive the standard of care for hyponatremia. Examples of the standard of care include limiting your water and fluid intake, or giving you salt tablets and other drugs such as diuretics. Your doctor will describe these in more detail.

You will be given a drug diary to record when you take the study drug/placebo. You will return any unused drug/placebo at the end of 14 days.

You should avoid grapefruit and grapefruit juice while you are taking tolvaptan.

Study Visits:

At every visit, you will be asked if you have had any side effects.

On Days 1, 2, and 3:

* Blood (about 1 teaspoon) will be drawn for routine tests. On Day 1, this sample will be drawn 2 times.
* Your weight and vital signs will be measured.
* The study staff will record how much fluid you are drinking and how much you are urinating.
* You will be asked about any drugs that you may be taking.
* If the doctor thinks it is needed, you will have a physical exam.

On Day 7:

* Your medical history will be reviewed and updated.
* You will be asked about any drugs that you may be taking.
* Blood (about 1 teaspoon) will be drawn for routine tests and tests to measure how concentrated your blood results are.
* Your weight and vital signs will be measured.

On Day 14:

* Your medical history will be reviewed and updated.
* Your weight and vital signs will be measured.
* Blood (about 1 teaspoon) and urine will be collected for routine tests and tests to measure how concentrated your blood and urine are.
* The study staff will record how much fluid you are drinking and how much you are urinating.
* You will be asked about any drugs that you may be taking.
* You will complete the MMSE.

If the doctor thinks it is needed, you will have a physical exam.

Length of Study:

You will take the study drug/placebo for 14 days. You will be taken off study if you have intolerable side effects, if the disease gets worse, or if the study doctor thinks it is in your best interest.

Your participation on the study will be over once you have completed the end-of-study visit.

End-of-Study- Day 30 Follow-up Visit:

At 30 days after the last dose of study drug (or placebo), you will have an end-of-study visit in clinic or by telephone. At this visit, the following tests and procedures will be performed.

* Your medical history will be reviewed and updated.
* Blood (about 1 teaspoon) will be drawn for routine tests and tests to measure how concentrated your blood results are.
* You will be asked about any side effects that you may be having and any drugs that you may be taking.
* The study staff will record how much fluid you are drinking and how much you are urinating.
* If the doctor thinks it is needed, you will have a physical exam.

This is an investigational study. Tolvaptan is FDA approved and commercially available to treat hyponatremia (low levels of salt [sodium] in the blood due to too much body water). Its use in patients with cancer who have hyponatremia is investigational.

Up to 170 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Euvolemic or hypervolemic (patients with heart or liver failure) with cancer admitted to MD Anderson Cancer Center for any reasons with serum sodium between 125 and 130 mEq/L (both inclusive)
2. Patients must be greater than or equal to 18 years of age
3. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3 at baseline.
4. Women of childbearing potential must use a medically accepted method of contraception and to continue use of this method for the duration of the study and for 30 days after study participation. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method. Men must practice abstinence or use a barrier method of birth control, and must agree to continue use for the duration of the study and for 30 days after study participation.
5. Subjects must be able to comply with scheduled visits and follow-ups.
6. Informed consent must be signed

Exclusion Criteria:

1. History of hypersensitivity to tolvaptan
2. Patients admitted to the critical care unit.
3. Patients with renal failure(creatinine clearance less than 25 ml/min)
4. Patients with a life expectancy less than 3 months
5. Patients with volume depletion, BP < 100/60 or urinary sodium <20 meq/L.
6. Patients who are not able to swallow or cannot take medication through feeding tubes
7. Patients with diuretic-induced hyponatremia.
8. Patients with spurious hyponatremia
9. Patients with hyponatremia related to psychogenic polydypsia, head trauma, post operative conditions, uncontrolled hypothyroidism or cortisol insufficiency or any hyponatremia associated with the use of medication that can be safely withdrawn.
10. The use of alcohol while participating in the study
11. Currently taking demeclocycline, lithium, benzazepine derivatives, ketoconazole, grapefruit, grapefruit juice and receiving strong CYP3A inhibitors such as clarithromycin, fluconazole, voriconazole, posaconazole, itraconazole, ritonavir, indinavir, nelfinavir, saquinavir, nefazodone, and telithromycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdulla K. Salahudeen, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 5, 2011 to July 13, 2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 52 participants enrolled, only 48 patients were randomized to participate in the study. Two participants were not randomized due to contra indicated medication and another two were not randomized due to exclusion criteria. The study was stopped for superiority.
Groups:
- Tolvaptan Group: Starting dose 15 mg orally once a day for 14 days.
- Placebo Group: Placebo orally once a day for 14 days.
Period: Overall Study
Arm/Group | Tolvaptan Group | Placebo Group
Started | 24 | 24
Completed | 17 | 13
Not Completed | 7 | 11
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 1 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — ICU Transfer | 1 | 2
Not completed — Hospice-care transfer | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline demographics and clinical characteristics of patients in the placebo group and the Tolvaptan Group who completed the 14-Day study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan Group | Placebo Group | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 60] | 69 [52 to 81] | 65 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Participants Whose Serum Sodium Concentration Corrected to at Least 135 mEq/L on Day 14
Description: Compare proportion of hyponatremia cancer patients with a normalized serum sodium concentration at day 14 between those treated with Tolvaptan and those treated with a placebo (standard of care). Proportion of participants whose serum sodium concentration is corrected to at least 136 mEq/Lon day14.
Time Frame: 14 days
Population: "Evaluable participants" are defined as all participants excluding those who drop out of the study due to non-study related reasons. Participants who are lost to follow-up for unknown or study related reasons will be counted as failures based on the intent to treat principal.
Measure: Number; unit: participants
Arm/Group | Tolvaptan Group | Placebo Group
Number analyzed (Participants) | 17 | 13
participants | 16 | 1

2. Secondary Outcome: Length of Stay in Hospital
Time Frame: From administration of treatment to time of discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tolvaptan Group | Placebo Group
Number analyzed (Participants) | 17 | 13
days | 21 (15) | 26 (15)

ADVERSE EVENTS:
Time Frame: Adverse event collection through follow up, anticipated Day 30 +/- 5 days. Overall collection period: May 10, 2011 to August 24, 2012.
Arm/Group | Tolvaptan Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 17/17 | 0/13
Other Adverse Events (participants affected / at risk) | 0/17 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan Group (N=17) | Placebo Group (N=13)
Pain (General disorders) | 17 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Edema (Skin and subcutaneous tissue disorders) | 17 | 0
Infections (any type) (Infections and infestations) | 13 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Hypotension (General disorders) | 8 | 0
Worsening of Edema (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes